CLINICAL TRIAL: NCT00499252
Title: A Phase II Evaluation of Abraxane® in the Treatment of Recurrent or Persistent Platinum-Resistant Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Brief Title: Paclitaxel Albumin-Stabilized Nanoparticle Formulation in Treating Patients With Recurrent or Persistent Ovarian Epithelial Cancer, Fallopian Tube Cancer, or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOG-0126R; NCI-2009-00575 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ABRAXIS-ABX-005; CDR0000553208; GOG-0126R (Other: Gynecologic Oncology Group); GOG-0126R (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2007-07-10; First posted 2007-07-11 (Estimated); Results first posted 2013-12-13 (Estimated); Last update posted 2018-01-11 (Actual); Status verified 2015-03

CONDITIONS: Fallopian Tube Carcinoma; Primary Peritoneal Carcinoma; Recurrent Ovarian Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Taxes; Albumin-Bound Paclitaxel

ARMS (1):
- Treatment (paclitaxel albumin-stabilized nanoparticle) (Experimental): Patients receive paclitaxel albumin-stabilized nanoparticle formulation (Abraxane®) IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Paclitaxel Albumin-Stabilized Nanoparticle Formulation

INTERVENTIONS:
Drug: Paclitaxel Albumin-Stabilized Nanoparticle Formulation
  Other Names: ABI 007; ABI-007; Abraxane

SUMMARY:
This phase II trial is studying the side effects and how well paclitaxel albumin-stabilized nanoparticle formulation works in treating patients with recurrent or persistent ovarian epithelial cancer, fallopian tube cancer, or primary peritoneal cancer. Drugs used in chemotherapy, such as paclitaxel albumin-stabilized nanoparticle formulation, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the antitumor activity of paclitaxel albumin-stabilized nanoparticle formulation (Abraxane®), in terms of frequency and duration of objective response, in patients with persistent or recurrent platinum-resistant ovarian epithelial, fallopian tube, or primary peritoneal cancer.

II. Determine the toxicity of this drug in these patients.

SECONDARY OBJECTIVES:

I. Determine the duration of progression-free survival and overall survival of patients treated with this drug.

OUTLINE: This is a multicenter study.

Patients receive paclitaxel albumin-stabilized nanoparticle formulation (Abraxane®) IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of 1 of the following:

  * Ovarian epithelial cancer
  * Fallopian tube cancer
  * Primary peritoneal carcinoma
* Recurrent or persistent disease
* Must have received 1 prior platinum-based chemotherapy regimen containing carboplatin, cisplatin, or another organoplatinum compound for management of primary disease

  * Initial treatment may have included intraperitoneal therapy, high-dose therapy, consolidation therapy, or extended therapy administered after a surgical or nonsurgical assessment
  * Patients who have not received prior paclitaxel-based chemotherapy must receive a second regimen that includes paclitaxel or docetaxel
* Platinum-resistant or refractory disease, defined by 1 of the following:

  * Treatment-free interval of < 6 months after completion of platinum-based therapy
  * Persistent disease at completion of primary platinum-based therapy
  * Progressive disease during platinum-based therapy
* Paclitaxel-resistant disease, defined as having had a treatment-free interval < 6 months or shown disease progression during paclitaxel-based therapy

  * Patients who have not received prior paclitaxel-based chemotherapy must receive a second regimen that includes paclitaxel or docetaxel
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques or ≥ 10 mm by spiral CT scan
* Must have ≥ 1 target lesion that can be used to assess response

  * Tumors within a previously irradiated field are designated as non-target lesions unless progression is documented or biopsy confirms persistence ≥ 90 days after completion of radiotherapy
* Not a candidate for a higher priority GOG protocol
* GOG performance status 0-2
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9.0 g/dL
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* Bilirubin normal
* SGOT ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN
* No active infection requiring antibiotics
* No sensory or motor neuropathy > grade 1
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* PT INR ≤ 1.5 or in-range INR 2-3 (if patient is on a stable dose of therapeutic warfarin)
* PTT < 1.2 times control
* No concurrent serious medical or psychiatric illness, including serious active infection
* No uncontrolled hypertension (i.e., blood pressure ≥ 150/100 mm Hg)
* No uncompensated congestive heart failure or symptomatic coronary artery disease
* No myocardial infarction within the past 6 months
* No active bleeding
* No other invasive malignancies within the past 5 years except for nonmelanoma skin cancer
* No history of allergic reactions attributed to chemical or biological composition to paclitaxel or other study agents
* No concurrent amifostine or other protective reagents
* Recovered from prior surgery, radiotherapy, or chemotherapy
* No prior paclitaxel albumin-stabilized nanoparticle formulation (Abraxane®)
* No prior cancer treatment that would preclude study therapy
* No additional prior cytotoxic chemotherapy for management of recurrent or persistent disease, including retreatment with initial chemotherapy regimens
* One additional prior noncytotoxic regimen (i.e., monoclonal antibodies, cytokines, or small molecule inhibitors of signal transduction) for management of recurrent or persistent disease allowed
* At least 1 week since prior hormonal therapy directed at the malignant tumor

  * Concurrent hormone replacement therapy allowed
* At least 3 weeks since other prior therapy directed at the malignant tumor, including biologic therapy, immunologic agents, or radiotherapy
* More than 5 years since prior chemotherapy for any other portion of the abdominal cavity or pelvis, unless for treatment of ovarian, primary peritoneal, or fallopian tube cancer

  * Prior adjuvant chemotherapy for localized breast cancer allowed provided it was completed > 3 years ago and patient remains free of recurrent or metastatic disease
* More than 5 years since prior radiotherapy to any other portion of the abdominal cavity or pelvis, unless for treatment of ovarian, primary peritoneal, or fallopian tube cancer

  * Prior radiotherapy for localized breast cancer, cancer of the head and neck, or skin cancer allowed provided it was completed > 3 years ago and patient remains free of recurrent or metastatic disease
* No prior radiotherapy to > 25% of marrow-bearing areas

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2007-06; Primary Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Coleman, Principal Investigator — Gynecologic Oncology Group
Locations (20):
- United States (20):
  - Colorado Gynecologic Oncology Group, Aurora, Colorado
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Rush University Medical Center, Chicago, Illinois
  - Union Hospital of Cecil County, Elkton, Maryland
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Roswell Park Cancer Institute, Buffalo, New York
  - North Shore University Hospital, Manhasset, New York
  - North Shore-LIJ Health System CCOP, Manhasset, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Riverside Methodist Hospital, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Cancer Care Associates-Midtown, Tulsa, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - University of Texas Medical Branch at Galveston, Galveston, Texas
  - Carilion Clinic Gynecological Oncology, Roanoke, Virginia
  - University of Washington Medical Center, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on 6/4/2007 and closed to accrual on 1/29/2009.
Groups:
- Abraxane®: Abraxane® 100 mg/m2 infused I.V. over 30 minutes weekly on days 1, 8, and 15 every 28 days until disease progression or adverse effects prohibit further therapy.
Period: Overall Study
Arm/Group | Abraxane®
Started | 51
Completed | 39 (Patients treated until disease progression; completed defined as off treatment due to progression.)
Not Completed | 12
Not completed — Adverse Event | 3
Not completed — Refused further treatment | 2
Not completed — Ineligible | 4
Not completed — <no further label> | 3

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients
Arm/Group | Abraxane®
Number analyzed (Participants) | 47
Age, Customized [Number; unit: participants]
  20-29 years | 0
  30-39 years | 1
  40-49 years | 8
  50-59 years | 16
  60-69 years | 15
  70-79 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response
Description: Complete and Partial Tumor Response by Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0). Per RECIST v1.0 for target lesions and assessed by MRIor CT scan: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest dimensions (LD) of all target measurable lesions taking as reference the baseline sum of LD.
  CT scan or MRI if used to follow lesion for measurable disease every other cycle for the first 6 months; every three months thereafter; and at any time if clinically indicated based on symptoms or physical signs suggestive of progressive disease or rising serum tumor marker levels. Responses must be confirmed by repeat imaging 4 weeks following documentation of response.
Time Frame: every other cycle for the first 6 months; every three months thereafter; and at any time if clinically indicated based on symptoms or physical signs suggestive of progressive disease or rising serum tumor marker levels
Population: Eligible and Treated Patients
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abraxane®
Number analyzed (Participants) | 47
Percentage of participants | 23.4 [12.3 to 38.0]

2. Primary Outcome: Frequency and Severity of Observed Adverse Effects
Time Frame: Every cycle during treatment and up to 5 years after completion of treatment
Population: Treated and Eligible patients
Measure: Count of Participants; unit: Participants
Groups:
- Grade 0: Number of patients who did not experience the specified AE.
- Grade 1 (CTCAE v 3.0): Number of patients who experienced a grade 1 event using Common Terminology Criteria version 3.0
- Grade 2 (CTCAE v 3.0): Number of patients who experienced a grade 2 event using Common Terminology Criteria version 3.0
- Grade 3 (CTCAE v 3.0): Number of patients who experienced a grade 3 event using Common Terminology Criteria version 3.0
Arm/Group | Grade 0 | Grade 1 (CTCAE v 3.0) | Grade 2 (CTCAE v 3.0) | Grade 3 (CTCAE v 3.0)
Number analyzed (Participants) | 47 | 47 | 47 | 47
Participants
  Leukopenia | 20 | 15 | 11 | 1
  Thrombocytopenia | 43 | 4 | 0 | 0
  Neutropenia | 30 | 5 | 6 | 6
  Anemia | 5 | 19 | 20 | 3
  Cardiac | 45 | 2 | 0 | 0
  Constitutional | 12 | 20 | 15 | 0
  Dermatologic | 28 | 10 | 9 | 0
  Gastrointestinal | 18 | 19 | 8 | 2
  Hemorrhage | 45 | 1 | 1 | 0
  Lymphatics | 41 | 6 | 0 | 0
  Metabolic | 35 | 8 | 2 | 2
  Musculoskeletal | 44 | 2 | 1 | 0
  Neurosensory | 27 | 14 | 5 | 1
  Other neurological | 42 | 4 | 1 | 0
  Ocular/Visual | 45 | 1 | 1 | 0
  Pain | 32 | 10 | 3 | 2
  Pulmonary | 40 | 3 | 4 | 0

3. Secondary Outcome: Progression-free Survival
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since study entry, or unequivocal progression of existing non-target lesions, or the appearance of one or more new lesions.
  CT scan or MRI if used to follow lesion for measurable disease every other cycle for the first 6 months; every three months thereafter; and at any time if clinically indicated based on symptoms or physical signs suggestive of progressive disease or rising serum tumor marker levels. Responses must be confirmed by repeat imaging 4 weeks following documentation of response.
Time Frame: from study entry until disease progression, death or date of last contact.
Population: Eligible and Treated Patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Abraxane®
Number analyzed (Participants) | 47
months | 4.5 [2.2 to 6.7]

4. Secondary Outcome: Overall Survival
Time Frame: from entry into the study to death or the date of last contact.
Population: Eligible and Treated Patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Abraxane®
Number analyzed (Participants) | 47
months | 17.4 [13.2 to 20.8]

ADVERSE EVENTS:
Time Frame: every cycle
Description: "Number of participants at risk" total includes eligible and treated patients.
Arm/Group | Abraxane®
Serious Adverse Events (participants affected / at risk) | 11/47
Other Adverse Events (participants affected / at risk) | 47/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abraxane® (N=47)
Ileus (Gastrointestinal disorders) | 2
Obstruction, Gi - Small Bowel Nos (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 1
Dehydration (Gastrointestinal disorders) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Skin(Cellulitis) (Infections and infestations) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Pain: Extremity-Limb (General disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Obstruction, Gu - Ureter (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abraxane® (N=47)
Rhinitis (Immune system disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Neutrophils (Blood and lymphatic system disorders) | 17
Platelets (Blood and lymphatic system disorders) | 4
Leukocytes (Blood and lymphatic system disorders) | 28
Hemoglobin (Blood and lymphatic system disorders) | 42
Palpitations (Cardiac disorders) | 1
Ventricular Arrhythmia - Tachycardia (Cardiac disorders) | 1
Hypertension (Cardiac disorders) | 1
Cardiac General - Other (Cardiac disorders) | 1
Hypotension (Cardiac disorders) | 1
Sweating (General disorders) | 1
Weight Gain (General disorders) | 5
Fever (General disorders) | 2
Weight Loss (General disorders) | 2
Rigors/Chills (General disorders) | 1
Fatigue (General disorders) | 33
Insomnia (General disorders) | 2
Nail Changes (Skin and subcutaneous tissue disorders) | 3
Photosensitivity (Skin and subcutaneous tissue disorders) | 1
Hair Loss/Alopecia (Scalp Or Body) (Skin and subcutaneous tissue disorders) | 19
Bruising (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 7
Dry Skin (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Hot Flashes (Endocrine disorders) | 3
Fistula, Gi - Small Bowel Nos (Gastrointestinal disorders) | 1
Esophagitis (Gastrointestinal disorders) | 1
Heartburn (Gastrointestinal disorders) | 3
Dental: Teeth (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Distention (Gastrointestinal disorders) | 3
Taste Alteration (Gastrointestinal disorders) | 2
Mucositis (Functional/Sympt) - Oral Cavity (Gastrointestinal disorders) | 2
Obstruction, Gi - Small Bowel Nos (Gastrointestinal disorders) | 3
Mucositis (Clinical Exam) - Oral Cavity (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 14
Anorexia (Gastrointestinal disorders) | 7
Dehydration (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 12
Nausea (Gastrointestinal disorders) | 21
Diarrhea (Gastrointestinal disorders) | 12
Hemorrhage, Gi - Rectum (Vascular disorders) | 1
Hemorrhage/Pulmonary - Nose (Vascular disorders) | 3
Hematoma (Vascular disorders) | 1
Petechiae (Vascular disorders) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Upper Airway Nos (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Oral Cavity-Gums (Infections and infestations) | 1
Inf Unknown Anc: Sinus (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Urinary Tract Nos (Infections and infestations) | 4
Inf W/Nml Or Gr 1 Or 2 Anc: Bronchus (Infections and infestations) | 1
Inf Unknown Anc: Upper Airway Nos (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Sinus (Infections and infestations) | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Bladder (Infections and infestations) | 2
Lymphedema-Related Fibrosis (Blood and lymphatic system disorders) | 1
Edema: Trunk/Genital (Blood and lymphatic system disorders) | 2
Edema: Limb (Blood and lymphatic system disorders) | 8
Ast (Metabolism and nutrition disorders) | 2
Creatinine (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Alt (Metabolism and nutrition disorders) | 2
Alkaline Phosphatase (Metabolism and nutrition disorders) | 2
Bilirubin (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 4
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 4
Hyperkalemia (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 6
Hypokalemia (Metabolism and nutrition disorders) | 4
Hypercalcemia (Metabolism and nutrition disorders) | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 7
Joint-Function (Musculoskeletal and connective tissue disorders) | 1
Joint Effusion (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Muscle Weakness - Whole Body/Generalized (Musculoskeletal and connective tissue disorders) | 1
Muscle Weakness - Extremity-Lower (Musculoskeletal and connective tissue disorders) | 1
Syncope (Nervous system disorders) | 1
Mood Alteration - Depression (Nervous system disorders) | 5
Mood Alteration - Anxiety (Nervous system disorders) | 5
Ataxia (Nervous system disorders) | 1
Memory Impairment (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 3
Neuropathy-Sensory (Nervous system disorders) | 24
Neuropathy-Motor (Nervous system disorders) | 3
Blurred Vision (Eye disorders) | 3
Pain - Other (General disorders) | 1
Pain: Pelvis (General disorders) | 1
Pain: Chest /Thorax Nos (General disorders) | 2
Pain: Head/Headache (General disorders) | 6
Pain: Extremity-Limb (General disorders) | 4
Pain: Buttock (General disorders) | 1
Pain: Back (General disorders) | 5
Pain: Joint (General disorders) | 7
Pain: Bone (General disorders) | 1
Pain: Pain Nos (General disorders) | 1
Pain: Stomach (General disorders) | 1
Pain: Rectum (General disorders) | 1
Pain: Abdominal Pain Nos (General disorders) | 14
Pain: Tumor (General disorders) | 1
Pain: Muscle (General disorders) | 1
Pain: Neuralgia (General disorders) | 1
Pulmonary: Other (Respiratory, thoracic and mediastinal disorders) | 3
Nasal/Paranasal Reactions (Respiratory, thoracic and mediastinal disorders) | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 11
Cystitis (Renal and urinary disorders) | 1
Incontinence, Urinary (Renal and urinary disorders) | 1
Urinary Frequency (Renal and urinary disorders) | 1
Vaginitis (Reproductive system and breast disorders) | 1
Vaginal Discharge (Reproductive system and breast disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No